CLINICAL TRIAL: NCT05701475
Title: Triple Prevention Against Cutibacterium Acnes Using Benzoyl Peroxide Preparation in Addition to Pre-operative Cutaneous and Subcutaneous Iodine in Shoulder Surgery; a Single-blinded, Randomized, Controlled Trial.
Brief Title: Cutibacterium Acnes: Triple Prevention in Shoulder Operations
Acronym: C3PO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Générale dAnnecy (Other)
Collaborators: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023C3PO-trial
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Post-Operative Wound Infection; Surgical Site Infection
Keywords: Cutibacterium Acnes; Prevention; Benzoyl peroxide; Subcutaneous disinfection; Surgical site infection; Pre-operative disinfection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Since the disinfection protocol has to be performed by the patient and care provider, this can not be blinded. However, the laboratory staff will not know which treatment arm the patient was allocated to when assessing the bacterial cultures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control/Single prevention (No Intervention): Standard pre-operative cutaneous disinfection using iodine.
- Double prevention (Experimental): Pre-operative cutaneous and subcutaneous disinfection using iodine.
  Interventions: Procedure: Subcutaneous disinfection
- Triple prevention (Experimental): Pre-operative cutaneous and subcutaneous disinfection using iodine and preparation of the skin with benzoyl peroxide in the days prior to surgery.
  Interventions: Procedure: Subcutaneous disinfection; Procedure: Benzoyl peroxide preparation

INTERVENTIONS:
Procedure: Subcutaneous disinfection — After incision, the subcutaneous tissue will be disinfected for 60 seconds using iodine before continuing the surgical approach.
  Arms: Double prevention; Triple prevention
Procedure: Benzoyl peroxide preparation — In the days prior to surgery, the skin will be prepared using Benzoyl Peroxide gel according to a standardised protocol.
  Arms: Triple prevention

SUMMARY:
Patients planned for shoulder surgery will be identified and contacted for participation. After informed consent is provided, patients will be randomised into one of three groups: pre-operative cutaneous disinfection with iodine (control group), pre-operative cutaneous and subcutaneous disinfection with iodine (double prevention), and pre-operative cutaneous and subcutaneous disinfection with iodine combined with a skin preparation protocol with benzoyl peroxide gel in the days prior to surgery (triple prevention). Bacterial cultures will be collected during surgery of the surgical field and tissue layers. Culture positivity for Cutibacterium Acnes will be compared between the groups as a primary outcome.

DETAILED DESCRIPTION:
Eligible patients will be contacted for participation (see Eligibility Criteria). If subjects meet the inclusion criteria, patients will receive information regarding the study outline, associated risks, and subject rights. Informed consent must be freely given, specific, unambiguous, and may be withdrawn at any time. Subjects must be legally capable of providing consent. Consent will be and recorded in writing and stored for the duration of the study. The target for inclusion was set at 52 patients in each group, of each group 26 will be arthroscopic and 26 open surgery.

Patients will be divided into three groups of equal size:

* Triple-prevention: Benzoyl peroxide at home, subcutaneous iodine, and cutaneous iodine.
* Double-prevention: Cutaneous and subcutaneous iodine.
* Single-prevention (control group): cutaneous iodine.

Simple block randomisation will be used to prevent chronological bias and ensure equal group size. Treatments will be allocated with a 1:1:1 ratio using a block size of 12. Randomisation will be stratified by open or arthroscopic surgery to ensure an equal number in all three groups (3x2x26 patients) Random treatment allocation numbers will be generated and blinded, to be revealed after inclusion.

Benzoyl peroxide:

Patients will be instructed to apply and rub in a 5-cm strip of 5% benzoyl peroxide gel to the shoulder on dry skin in the morning and evening 2 days prior to surgery, 1 day before surgery, and a fifth time in the morning on the day of surgery.

Cutaneous iodine:

Standard pre-operative preparation including cutaneous disinfection with alcoholic iodine, sterile drapes.

Subcutaneous iodine:

Open surgery: after incision down to the fascia of the muscle layer, preparation of the whole subcutaneous layer with povidone-iodine solution will be performed and left acting during 60 seconds before full aspiration and lavage in order to not have swabs drained in povidone-iode (as it could continue to act as antiseptic during culture).

For arthroscopic procedures the disinfection and swab collection protocol will be performed when creating the first portal.

Bacterial culture swabs (n=9) will be taken during surgery from the patients' skin (before disinfection with iodine), subcutaneous tissue (after disinfection if randomised for subcutaneous disinfection), muscular layer, intra-articular/layer of the intervention (for example in case of clavicle surgery from the clavicle), surgeon's glove, outside scalpel, inside scalpel, and the retractors. For the swabs in the operative field, the applicable field is to be swabbed fully for 3 seconds. Each surgeon will follow the clear swab instructions from the microbiologist in order to obtain reliable cultures. Cultures will be analysed by the hospital's medical microbiological laboratory following standard protocol including a standard incubation time of 14 days. Treatment arm will be blinded for the laboratory employees.

Culture positivity between the groups will be analysed using chi-square tests for each culture location. In addition, a two-way ANOVA test will be performed to assess total number of positive cultures per patient. Furthermore, logistic regression models will be used to adjust for several potential confounding factors depending on the number of positive tests in the sample.

ELIGIBILITY:
Inclusion Criteria:

* Indication for all types of surgery at the shoulder joint, acromioclavicular joint, or clavicle, including arthroscopic and open surgery.

Exclusion Criteria:

* Previous shoulder surgery;
* History of shoulder infection;
* Antibiotic treatment in the last 6 weeks;
* Allergy or hypersensitivity to one of the disinfecting agents;
* Patients with laboratory values consistent with a current infection (C-reactive protein, erythrocyte sedimentation rate, leukocyte count).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Cutibacterium Acnes positivity | 14 days
  Rate of culture positivity for Cutibacterium Acnes of swabs taken during surgery

SECONDARY OUTCOMES:
Culture positivity with other bacteria | 14 days
  Rate of culture positivity for other types of bacteria of swabs taken during surgery
Adherence to pre-operative protocol | 1 day
  Completeness percentage of the pre-operative skin preparation protocol as reported by participants the morning of the intervention

OTHER OUTCOMES:
Adverse reaction to Benzoyl Peroxide | 1 day
  Number and type of adverse reactions of any type to Benzoyl Peroxide reported by participants

CONTACTS AND LOCATIONS:
Overall Officials: Geert A Buijze, MD, PhD, Principal Investigator — Clinique Générale d'Annecy
Locations (1):
- Clinique Générale d'Annecy, Annecy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore NF, Batten TJ, Hutton CE, White WJ, Smith CD. The management of the shoulder skin microbiome (Cutibacterium acnes) in the context of shoulder surgery: a review of the current literature. Shoulder Elbow. 2021 Oct;13(6):592-599. doi: 10.1177/1758573220945226. Epub 2020 Jul 27. PMID 34804207
- [Background] Moor BK, Leger B, Steffen V, Troillet N, Emonet S, Gallusser N. Subcutaneous tissue disinfection significantly reduces Cutibacterium acnes burden in primary open shoulder surgery. J Shoulder Elbow Surg. 2021 Jul;30(7):1537-1543. doi: 10.1016/j.jse.2020.11.018. Epub 2021 Jan 6. PMID 33421560
- [Background] Kaveeshwar S, Duvall G, Jones DL, O'Hara NN, Klein A, Diedrich AM, Kolakowski L, Lai JK, Hasan SA, Henn RF 3rd, Gilotra MN. Risk factors for increased shoulder Cutibacterium acnes burden. JSES Int. 2020 Jun 3;4(3):464-469. doi: 10.1016/j.jseint.2020.04.020. eCollection 2020 Sep. PMID 32939469
- [Background] Hudek R, Brobeil A, Bruggemann H, Sommer F, Gattenlohner S, Gohlke F. Cutibacterium acnes is an intracellular and intra-articular commensal of the human shoulder joint. J Shoulder Elbow Surg. 2021 Jan;30(1):16-26. doi: 10.1016/j.jse.2020.04.020. Epub 2020 Jun 9. PMID 32741563
- [Background] Lavergne V, Malo M, Gaudelli C, Laprade M, Leduc S, Laflamme P, Rouleau DM. Clinical impact of positive Propionibacterium acnes cultures in orthopedic surgery. Orthop Traumatol Surg Res. 2017 Apr;103(2):307-314. doi: 10.1016/j.otsr.2016.12.005. Epub 2017 Jan 5. PMID 28065868
- [Background] Chalmers PN, Beck L, Stertz I, Tashjian RZ. Hydrogen peroxide skin preparation reduces Cutibacterium acnes in shoulder arthroplasty: a prospective, blinded, controlled trial. J Shoulder Elbow Surg. 2019 Aug;28(8):1554-1561. doi: 10.1016/j.jse.2019.03.038. Epub 2019 Jun 20. PMID 31229329
- [Background] Singh AM, Sethi PM, Romeo AA, Anakwenze OA, Abboud JA, Namdari S. Strategies to decolonize the shoulder of Cutibacterium acnes: a review of the literature. J Shoulder Elbow Surg. 2020 Apr;29(4):660-666. doi: 10.1016/j.jse.2019.11.037. PMID 32197761
- [Background] Dizay HH, Lau DG, Nottage WM. Benzoyl peroxide and clindamycin topical skin preparation decreases Propionibacterium acnes colonization in shoulder arthroscopy. J Shoulder Elbow Surg. 2017 Jul;26(7):1190-1195. doi: 10.1016/j.jse.2017.03.003. Epub 2017 May 4. PMID 28479255
- [Background] Kolakowski L, Lai JK, Duvall GT, Jauregui JJ, Dubina AG, Jones DL, Williams KM, Hasan SA, Henn RF 3rd, Gilotra MN. Neer Award 2018: Benzoyl peroxide effectively decreases preoperative Cutibacterium acnes shoulder burden: a prospective randomized controlled trial. J Shoulder Elbow Surg. 2018 Sep;27(9):1539-1544. doi: 10.1016/j.jse.2018.06.012. Epub 2018 Jul 24. PMID 30054245
- [Background] Sabetta JR, Rana VP, Vadasdi KB, Greene RT, Cunningham JG, Miller SR, Sethi PM. Efficacy of topical benzoyl peroxide on the reduction of Propionibacterium acnes during shoulder surgery. J Shoulder Elbow Surg. 2015 Jul;24(7):995-1004. doi: 10.1016/j.jse.2015.04.003. PMID 26067191
- [Background] Scheer VM, Bergman Jungestrom M, Lerm M, Serrander L, Kalen A. Topical benzoyl peroxide application on the shoulder reduces Propionibacterium acnes: a randomized study. J Shoulder Elbow Surg. 2018 Jun;27(6):957-961. doi: 10.1016/j.jse.2018.02.038. Epub 2018 Mar 30. PMID 29609999
- [Background] van Diek FM, Pruijn N, Spijkers KM, Mulder B, Kosse NM, Dorrestijn O. The presence of Cutibacterium acnes on the skin of the shoulder after the use of benzoyl peroxide: a placebo-controlled, double-blinded, randomized trial. J Shoulder Elbow Surg. 2020 Apr;29(4):768-774. doi: 10.1016/j.jse.2019.11.027. PMID 32197765
- [Background] Scheer VM, Jungestrom MB, Serrander L, Kalen A, Scheer JH. Benzoyl peroxide treatment decreases Cutibacterium acnes in shoulder surgery, from skin incision until wound closure. J Shoulder Elbow Surg. 2021 Jun;30(6):1316-1323. doi: 10.1016/j.jse.2020.12.019. Epub 2021 Feb 3. PMID 33545336
- [Background] Hsu JE, Whitson AJ, Woodhead BM, Napierala MA, Gong D, Matsen FA 3rd. Randomized controlled trial of chlorhexidine wash versus benzoyl peroxide soap for home surgical preparation: neither is effective in removing Cutibacterium from the skin of shoulder arthroplasty patients. Int Orthop. 2020 Jul;44(7):1325-1329. doi: 10.1007/s00264-020-04594-x. Epub 2020 May 8. PMID 32385554
- [Background] Green N, Jordan RW, Maclean S, D'Alessandro P, MacDonald PB, Malik SS. Preoperative topical benzoyl peroxide treatment is effective in reducing Cutibacterium acnes in shoulder surgery: a systematic review. J Shoulder Elbow Surg. 2023 Jan;32(1):213-222. doi: 10.1016/j.jse.2022.07.019. Epub 2022 Sep 5. PMID 36067940
- [Background] Stull JD, Nicholson TA, Davis DE, Namdari S. Addition of 3% hydrogen peroxide to standard skin preparation reduces Cutibacterium acnes-positive culture rate in shoulder surgery: a prospective randomized controlled trial. J Shoulder Elbow Surg. 2020 Feb;29(2):212-216. doi: 10.1016/j.jse.2019.09.038. Epub 2019 Dec 13. PMID 31839392
- [Background] Rao AJ, Chalmers PN, Cvetanovich GL, O'Brien MC, Newgren JM, Cole BJ, Verma NN, Nicholson GP, Romeo AA. Preoperative Doxycycline Does Not Reduce Propionibacterium acnes in Shoulder Arthroplasty. J Bone Joint Surg Am. 2018 Jun 6;100(11):958-964. doi: 10.2106/JBJS.17.00584. PMID 29870447
- [Background] Namdari S, Nicholson T, Parvizi J, Ramsey M. Preoperative doxycycline does not decolonize Propionibacterium acnes from the skin of the shoulder: a randomized controlled trial. J Shoulder Elbow Surg. 2017 Sep;26(9):1495-1499. doi: 10.1016/j.jse.2017.06.039. Epub 2017 Jul 19. PMID 28734717
- [Background] Matsen FA, Whitson AJ, Hsu JE. While home chlorhexidine washes prior to shoulder surgery lower skin loads of most bacteria, they are not effective against Cutibacterium (Propionibacterium). Int Orthop. 2020 Mar;44(3):531-534. doi: 10.1007/s00264-019-04477-w. Epub 2020 Jan 14. PMID 31938858
- [Background] MacLean SBM, Phadnis J, Ling CM, Bain GI. Application of dermal chlorhexidine antisepsis is ineffective at reducing Proprionibacterium acnes colonization in shoulder surgery. Shoulder Elbow. 2019 Apr;11(2):98-105. doi: 10.1177/1758573218755570. Epub 2018 Jan 30. PMID 30936948
- [Background] Duvall G, Kaveeshwar S, Sood A, Klein A, Williams K, Kolakowski L, Lai J, Enobun B, Hasan SA, Henn RF 3rd, Gilotra MN. Benzoyl peroxide use transiently decreases Cutibacterium acnes load on the shoulder. J Shoulder Elbow Surg. 2020 Apr;29(4):794-798. doi: 10.1016/j.jse.2019.06.026. Epub 2019 Oct 31. PMID 31676186